CLINICAL TRIAL: NCT02005042
Title: Developing a Real-time, Ecologically Sensitive Physical Activity Intervention Using Smartphones and Bluetooth-enabled Pedometers: Feasibility and Initial Efficacy
Brief Title: Physical Activity and Daily Experiences Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTSI-BENI-Heron
Record Dates: First submitted 2013-11-22; First posted 2013-12-09 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Physical Activity
Keywords: Physical activity; Ecological Momentary Assessment; Ecological Momentary Intervention; Accelerometer; Smartphone
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Accelerometer only (No Intervention): Wear accelerometer only to measure activity levels (steps)
- Accelerometer plus EMA (No Intervention): Wear accelerometer and complete Ecological Momentary Assessment (EMA) surveys on smartphone 5 times daily
- Feedback on smartphone (Experimental): Wear accelerometer, complete EMA surveys on smartphone 5 times daily, receive intervention
  Interventions: Behavioral: Feedback on smartphone

INTERVENTIONS:
Behavioral: Feedback on smartphone — Receive personalized feedback (EMI) on smartphone regarding physical activity
  Arms: Feedback on smartphone

SUMMARY:
Lack of physical activity is associated with negative health outcomes, including obesity, diabetes, and cardiovascular disease. There are calls from NIH and medical organizations to integrate the use mobile devices, such as smartphones, to provide "e-health" interventions to patients in their daily life. Referred to as Ecological Momentary Interventions [EMI], these innovative mobile methods provide an opportunity for researchers and clinicians to offer tailored intervention material to people at specific times and in specific settings when they may be most in need of such support. To our knowledge no study has used objective ambulatory assessment data to deliver EMI. This preliminary work is to demonstrate the feasibility, and test preliminary efficacy, of using a Bluetooth accelerometer to provide real-time feedback on a smartphone to increase objectively measured steps (i.e., increase activity). A within-person design will be used, including assessment, intervention, and follow-up phases. During the assessment phase objective physical activity (using accelerometers) will be collected. In the intervention phase participants will also receive real-time feedback throughout the day regarding their total steps and personalized step goals. Objectively measured steps and disease status measures will be used to evaluate efficacy.

DETAILED DESCRIPTION:
Lack of physical activity is associated with negative health outcomes, including obesity, diabetes, and cardiovascular disease. A myriad of interventions aimed at increasing daily physical activity (PA) exist. Increasing PA levels has been shown to improve health among patients with cardiovascular and metabolic diseases. Accelerometers and pedometers can be useful tools in such interventions, particularly when used to provide participants with individualized feedback on progress toward PA goals. These programs typically require participants to set PA goals (e.g., number of steps/day), wear pedometers, and record daily activity levels from the pedometers. This process relies heavily on accurate self-reported information and is both time- and effort-intensive for participants, thus limiting acceptability and longer-term viability of this intervention option.

There is an increasing trend in health behavior research to use mobile devices, such as smartphones to provide interventions. These methods - known as Ecological Momentary Interventions [EMI] - are innovative because they allow researchers and clinicians to offered information to people at specific times and in settings when they may be most in need of such support. One way EMI can be tailored is by having participants complete repeated self-report assessments on mobile devices such as smartphones (known as Ecological Momentary Assessment [EMA]), and then using this material to identify times when people are in need of intervention. Although some studies (including recent studies conducted by members of our research team) have developed interventions that use EMA to create real-time interventions that are delivered in daily life, to our knowledge no study has used objective ambulatory assessment data to do so. Using objective data is potentially advantageous because it utilizes passive data collection (requiring little or no input by participants), and thus reduces participant burden and potential concerns regarding accuracy of self-reported data.

The first aim of this study is to establish the feasibility and acceptability of integrating Bluetooth-enabled activity monitor with smartphones to provide real-time feedback regarding physical activity in everyday life. We will evaluate feasibility and acceptability of this intervention method by tracking intervention delivery and participant compliance with EMA. This information will be automatically recorded by smartphone and activity monitor.

The second aim of this work is to provide a preliminary evaluation of the efficacy of delivering real-time feedback based on objectively measured PA. Our primary outcome is number of objectively measured steps. It is expected that participants will increase from their baseline number of steps when receiving personalized feedback and reminders on the smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English literate
* A BMI ranging from 25-40 (overweight or obese), based on self-report height and weight
* Not meeting current national physical activity guidelines
* Self-report they are able to walk unassisted, without the help of a wheel chair, walker, cane, crutches, or other walking aids
* Medically cleared to participate by completing screening form
* For women: not currently pregnant or actively trying to get pregnant for duration of study

Exclusion Criteria:

* Younger than 18
* Not English literate
* Self-report they are unable to walk unassisted, without the help of a wheel chair, walker, cane, crutches, or other walking aids
* A BMI outside of inclusion range (<25 or >40), based on self-report height and weight
* Meeting current national physical activity guidelines
* Not medically cleared to participate
* For women: currently pregnant or actively trying to get pregnant for duration of study. Pregnant women or those trying to become pregnant will be excluded because pregnancy may interfere with women's ability to go about previously normal activities, and will influence our outcome measures (e.g., BMI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of steps | during intervention (~28 days)

SECONDARY OUTCOMES:
BMI | Baseline, Post-intervention
blood pressure | Baseline
Hemoglobin A1c | Baseline
waist-hip ratio | Baseline

OTHER OUTCOMES:
Perceived Stress | Baseline, Post-intervention
  Perceived Stress Scale
Depression | Baseline, Post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D)
Social Support | Baseline, Post-intervention
  Social Network Index Survey
Satisfaction with Life | Baseline, Post-intervention
  Satisfaction with Life Scale
Barriers for Physical Activity | Baseline, Post-intervention
  Barriers for Physical Activity Questionnaire
Social Support and Exercise | Baseline, Post-intervention
  Social Support and Exercise Survey
Outcomes of Exercise | Baseline, Post-intervention
  Outcomes of Exercise Questionnaire
Walking measure | Baseline, Post-intervention
  Walking Questionnaire
Habit Index for Physical Activity | Baseline, Post-intervention
  Habit Index for Physical Activity
Rumination | Baseline, Post-intervention
  Rumination Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Heron, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States